CLINICAL TRIAL: NCT05447104
Title: Assessment of Salivary Flow Promoted by Sugar-Free Chewing Gum in Healthy Adults
Brief Title: Salivary Flow Promoted by Sugar-Free Chewing Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mars Wrigley (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M.WRI-2021-SAL-03
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Saliva Altered
Keywords: "salivary flow rate", saliva
MeSH Terms: interventions — Mastication

STUDY DESIGN:
Intervention Model Description: prospectively planned, double-blind, single center cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADA Clinically-Tested Reference Sugar-Free Gum (Active Comparator): Peppermint flavored sugar-free chewing gum (1 piece = 2.2 grams)
  Interventions: Behavioral: Mastication
- Marketed Gum: Sugar-free gum (Experimental): Orbit White, peppermint flavored sugar-free chewing gum Mars Wrigley Confectionary US, LLC (1 piece = 2.0 grams)
  Interventions: Behavioral: Mastication

INTERVENTIONS:
Behavioral: Mastication — Chewing sugar-free gum for 20 min

SUMMARY:
This was a double-blind, single center in vivo salivary flow rate study. The objective was to compare a marketed sugar-free chewing gum to a clinically-tested sugar-free reference chewing gum, with regards to their ability to promote salivary flow during a 20-minute chew period in healthy human adult subjects. Two sugar-free chewing gums were randomly assigned and distributed in a cross-over fashion to study subjects over two test period visits. The primary response being measured was salivary flow promoted by sugar-free chewing gums during the 20-minute chewing period.

DETAILED DESCRIPTION:
These procedures were conducted in accordance with proposed guidelines for current good clinical practices. Informed consent was obtained in compliance with FDA regulations (21 CFR 50). Each subject read, understood, signed, and received a signed copy of the most current IRB approved informed consent document prior to any study-related procedures being performed. The test and control gums were provided by the Sponsor. One serving size of each gum type was placed in a labeled, small high barrier foil bag to ensure that the subjects and the site personnel received the gum in a blinded manner. During each of the test visits, subjects: 1) provided a non-stimulated saliva sample to ensure continued qualification, 2) received their assigned chewing gum, and 3) provided stimulated saliva over a timed 20-minute chewing period. The primary response being measured was the salivary flow promoted by each chewing gum.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* have the ability to understand the information contained in the informed consent without the need for cognitive or language interpretation from any other person or source
* read, comprehend and sign the Informed Consent and other necessary paperwork prior to initiation of study procedures
* be in good general health based on his/her medical and dental history
* have a reasonably functional dentition with a minimum of 20 natural teeth (8 of which are posterior teeth)
* chew gum at least occasionally, no less than one time per month
* have normal salivary flow as demonstrated by being able to expectorate ≥ 1.5 mL (0.3 mL/min) of whole non-stimulated saliva over a 5-minute period
* be willing to participate in the study, be able to follow the study directions, and be willing to return for all specified visits at their appointed time, and
* be willing to postpone all elective dental procedures, at the Principal Investigator/Examiner's discretion, until the study has been completed.

Exclusion Criteria:

* advanced periodontal disease
* five or more grossly decayed, untreated dental sites (cavities)
* pathologic lesions of the oral cavity (suspicious or confirmed)
* full or partial dentures, or fixed orthodontic appliances, with the exception of a fixed, lower lingual retainer
* (if female) a medical history indicating that the subject is pregnant or currently breastfeeding
* current participation in another clinical research study or recent participation in another clinical trial (within 30 days of the study start date) may be cause for exclusion, based on the discretion of the Principal Investigator/Dental Examiner
* a history of a true allergy or intolerance to gum ingredients, including (but not limited to) sweeteners, colors or flavors, mint, peppermint, spearmint, milk proteins, or other ingredients which may be present in the study products
* Have a serious medical illness or disorder, e.g., immune compromised, AIDs, etc., that would be unduly affected by participation in this study, per the Principal Investigator/Dental Examiner's discretion
* a history of PKU (an intolerance to phenylalanine)
* a true food allergy to soy, or
* a history of temporomandibular disorder (TMD).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Salivary flow rate | 20 min
  Rate of healthy, adult human salivary flow rate while chewing sugar free gum

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Matis, Principal Investigator — Therametric Technologies, Inc.
Locations (1):
- Therametric Technologies, Inc., Noblesville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No